CLINICAL TRIAL: NCT03000478
Title: Virtual Reality Treatment for Combat Related PTSD: Is Virtual Azza More Effective Than Traditional Exposure Treatment?
Brief Title: Virtual Reality Exposure Therapy for Combat
Acronym: VRET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Sara Freedman, Dr. Sara Freedman, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIU201216
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure (Active Comparator): 12 sessions of PE as per protocol
  Interventions: Behavioral: Prolonged Exposure
- VRET (Experimental): 12 sessions of Virtual Reality Exposure Therapy
  Interventions: Behavioral: Virtual Reality Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure
  Arms: Prolonged Exposure
Behavioral: Virtual Reality Exposure Therapy
  Arms: VRET

SUMMARY:
This non inferiority trial will compare Prolonged Exposure with Virtual Reality Exposure Therapy in adult patients with combat related PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) affects a significant number of combat soldiers, with some studies suggesting 20% have PTSD. PTSD is related to a number of other detrimental effects, on the individual, such as mood disorders and alcohol abuse, on family members, and on society at large. Although effective treatments for PTSD exist, primarily types of cognitive behavior therapy, their uptake is very low. Studies have shown that a variety of factors act as barriers to care. These include not having the time for therapy, no therapy being locally available, and general stigma about therapy. In military populations, this stigma includes worries about the attitudes of unit members and commanding officers. As a result, many combat veterans do not seek therapy. Recently, it has been suggested that providing therapy in non-conventional settings might overcome some of these barriers. Studies over the last decade have shown that using Virtual Reality is a potential option. Virtual reality is a computer based environment that allows the therapist complete control over its multimedia components. VR is easily adaptable to exposure based treatments, where patients gradually come into contact with feared situations. VR for PTSD following combat, terror and motor vehicle accidents have all shown to be effective treatments. The studies so far are few, involve a small number of patients, and have often not adhered to gold standards of controlled trials. In addition, VR for combat in Israel has never been developed or tested.

The current study is a randomized controlled trial, that will compare traditional face-to-face treatment with Virtual Reality, for combat related PTSD. Blind assessors will examine levels of PTSD and other disorders before treatment, immediately after treatment, and at 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* combat related PTSD; Hebrew first language

Exclusion Criteria:

* suicidality, other psychiatric diagnosis requiring treatment, concurrent treatment,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms | 6 months post treatment
  PTSD as measured by the CAPS

CONTACTS AND LOCATIONS:
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No